CLINICAL TRIAL: NCT01082328
Title: ENDURE: A Phase IV, Prospective, Open-label, Uncontrolled, Multi-centre Cohort Trial to Assess the Responsiveness of Subjects With Phenylketonuria (PKU) to Treatment With Kuvan® 20 mg/kg/Day for 28 Days
Brief Title: Response to Kuvan® in Subjects With Phenylketonuria (PKU) in a 4 Weeks Testing Period
Acronym: ENDURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Norway (Industry); Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700773-503
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria (PKU); Hyperphenylalaninemia (HPA); Kuvan®; Sapropterin dihydrochloride; Kuvan responder; Tetrahydrobiopterin (BH4)
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kuvan® (Experimental)
  Interventions: Drug: Kuvan®

INTERVENTIONS:
Drug: Kuvan® — Kuvan® (sapropterin dihydrochloride) oral solution 20 milligram per kilogram (mg/kg) will be given once daily for 28 +/- 1 days.
  Other Names: Sapropterin dihydrochloride

SUMMARY:
The primary objective of the study is to evaluate the proportion of responders (that is, greater than or equal to [>=] 30 percent reduction from Baseline in blood phenylalanine [Phe] level) to treatment with Kuvan® (sapropterin dihydrochloride) 20 milligram per kilogram per day (mg/kg/day) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 4 years or older at the time the informed consent is obtained
* Subjects diagnosed with PKU (subgroups defined as: classic PKU [blood Phe greater than {>}1200 micromole per liter {mcmol/L}], mild PKU [blood Phe 600 to1200 mcmol/L] or mild hyperphenylalaninemia (HPA) [blood Phe 300 to 600 mcmol/L]
* Subjects who have received no previous treatment with sapropterin dihydrochloride (either Kuvan® or any other formulations of tetrahydrobiopterin [BH4])
* Subjects adherent to their normal diet and willing to adhere to the given diet for the 4 weeks study period
* Subjects who provide a signed (by parent if below 18 years) written informed consent
* Subjects with documented genotyping for both phenylalanine hydroxylase (PAH) mutations (PKU genotype)
* Phenylketonuria (PKU) diagnosis should be documented with at least two historical blood Phe levels above 400 mcmol/L
* Female subjects of childbearing potential (and, if appropriate, male subjects with female partners of childbearing potential) must be willing to avoid pregnancy by using an adequate method of contraception (defined as two barrier methods or one barrier method with spermicide, or intrauterine device or use of the oral female contraceptive) for 4 weeks prior to, during and 12 weeks after the last dose of trial medication
* Women of childbearing potential (for the purpose of this trial, women of childbearing potential are defined as "All female subjects after puberty unless they are post-menopausal for at least 2 years, are surgically sterile or are sexually inactive") must have a negative urine pregnancy test at the Baseline visit

Exclusion Criteria:

* Subjects who have documented BH4 deficiency
* Subjects who have any contraindications to receive Kuvan® as outlined in the summary of product characteristics (SmPC) not willing or able to comply with the study procedures
* Subjects who are pregnant, planning for pregnancy or breastfeeding
* Subjects who have been exposed to any investigational medicinal drugs or treatments within 30 days or 5 half-lives, whichever is longer, prior to the Screening visit
* Subjects using concomitant treatment with folate synthesis inhibiting drugs
* Subjects with concurrent use of Levodopa
* Subjects with concurrent use of inhibitors of dihydrofolate reductase (for example, methotrexate, trimethoprim)
* Subjects with concurrent use of agents that cause vasodilation, including those administered topically, by affecting nitric oxide (NO) metabolism or action including classical NO donors (for example, glyceryl trinitrate (GTN), isosorbide dinitrate (ISDN), sodium nitroprusside (SNP), molsidomin), phosphodiesterase type 5 (PDE-5) inhibitors and minoxidil
* Subjects who have a concurrent disease potentially interfering safety (for example, seizure disorder, oral steroid dependent asthma, other conditions requiring systemic corticosteroids, or insulin-dependent diabetes mellitus)
* Subjects who have inadequate liver function, defined by alanine aminotransferase (ALT) >= 2 times upper limit of normal (ULN)
* Subjects who have clinically significant renal dysfunction, defined by serum creatinine > 250 mcmol/L
* Have any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug or would significantly interfere with the subject's ability to comply with the provisions of the protocol

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Department of Paediatric Research, Division of Paediatrics, Oslo University Hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Scriver CR, Kaufman S. Hyperphenylanaemia: phenylalanine hydroxylase deficiency. In: Beaudet AL, Sly WS, Valle D, editors. Metabolic and molecular bases of inherited disease. New York: McGraw-Hill 2001;1667-709
- [Background] Phenylketonuria (PKU): screening and management. NIH Consens Statement. 2000 Oct 16-18;17(3):1-33. PMID 11757784
- [Background] Hofman KJ, Steel G, Kazazian HH, Valle D. Phenylketonuria in U.S. blacks: molecular analysis of the phenylalanine hydroxylase gene. Am J Hum Genet. 1991 Apr;48(4):791-8. PMID 2014802
- [Background] Konecki DS, Lichter-Konecki U. The phenylketonuria locus: current knowledge about alleles and mutations of the phenylalanine hydroxylase gene in various populations. Hum Genet. 1991 Aug;87(4):377-88. doi: 10.1007/BF00197152. PMID 1679029
- [Background] Kaufman S. An evaluation of the possible neurotoxicity of metabolites of phenylalanine. J Pediatr. 1989 May;114(5):895-900. doi: 10.1016/s0022-3476(89)80161-1. No abstract available. PMID 2654351
- [Background] Huttenlocher PR. The neuropathology of phenylketonuria: human and animal studies. Eur J Pediatr. 2000 Oct;159 Suppl 2:S102-6. doi: 10.1007/pl00014371. PMID 11043154
- [Background] Walter JH, White FJ, Hall SK, MacDonald A, Rylance G, Boneh A, Francis DE, Shortland GJ, Schmidt M, Vail A. How practical are recommendations for dietary control in phenylketonuria? Lancet. 2002 Jul 6;360(9326):55-7. doi: 10.1016/s0140-6736(02)09334-0. PMID 12114043
- [Background] Koch R, Azen C, Friedman EG, Williamson ML. Paired comparisons between early treated PKU children and their matched sibling controls on intelligence and school achievement test results at eight years of age. J Inherit Metab Dis. 1984;7(2):86-90. doi: 10.1007/BF01805813. PMID 6434835
- [Background] Brumm VL, Azen C, Moats RA, Stern AM, Broomand C, Nelson MD, Koch R. Neuropsychological outcome of subjects participating in the PKU adult collaborative study: a preliminary review. J Inherit Metab Dis. 2004;27(5):549-66. doi: 10.1023/b:boli.0000042985.02049.ff. PMID 15669671
- [Background] Kure S, Hou DC, Ohura T, Iwamoto H, Suzuki S, Sugiyama N, Sakamoto O, Fujii K, Matsubara Y, Narisawa K. Tetrahydrobiopterin-responsive phenylalanine hydroxylase deficiency. J Pediatr. 1999 Sep;135(3):375-8. doi: 10.1016/s0022-3476(99)70138-1. PMID 10484807
- [Background] Muntau AC, Roschinger W, Habich M, Demmelmair H, Hoffmann B, Sommerhoff CP, Roscher AA. Tetrahydrobiopterin as an alternative treatment for mild phenylketonuria. N Engl J Med. 2002 Dec 26;347(26):2122-32. doi: 10.1056/NEJMoa021654. PMID 12501224
- [Background] Trefz FK, Scheible D, Frauendienst-Egger G, Korall H, Blau N. Long-term treatment of patients with mild and classical phenylketonuria by tetrahydrobiopterin. Mol Genet Metab. 2005 Dec;86 Suppl 1:S75-80. doi: 10.1016/j.ymgme.2005.06.026. Epub 2005 Oct 20. PMID 16242984
- [Background] Shintaku H, Kure S, Ohura T, Okano Y, Ohwada M, Sugiyama N, Sakura N, Yoshida I, Yoshino M, Matsubara Y, Suzuki K, Aoki K, Kitagawa T. Long-term treatment and diagnosis of tetrahydrobiopterin-responsive hyperphenylalaninemia with a mutant phenylalanine hydroxylase gene. Pediatr Res. 2004 Mar;55(3):425-30. doi: 10.1203/01.PDR.0000111283.91564.7E. Epub 2003 Dec 17. PMID 14681498
- [Background] Hennermann JB, Buhrer C, Blau N, Vetter B, Monch E. Long-term treatment with tetrahydrobiopterin increases phenylalanine tolerance in children with severe phenotype of phenylketonuria. Mol Genet Metab. 2005 Dec;86 Suppl 1:S86-90. doi: 10.1016/j.ymgme.2005.05.013. Epub 2005 Jul 26. PMID 16051511
- [Background] Belanger-Quintana A, Garcia MJ, Castro M, Desviat LR, Perez B, Mejia B, Ugarte M, Martinez-Pardo M. Spanish BH4-responsive phenylalanine hydroxylase-deficient patients: evolution of seven patients on long-term treatment with tetrahydrobiopterin. Mol Genet Metab. 2005 Dec;86 Suppl 1:S61-6. doi: 10.1016/j.ymgme.2005.07.024. Epub 2005 Sep 13. PMID 16165389
- [Background] Lambruschini N, Perez-Duenas B, Vilaseca MA, Mas A, Artuch R, Gassio R, Gomez L, Gutierrez A, Campistol J. Clinical and nutritional evaluation of phenylketonuric patients on tetrahydrobiopterin monotherapy. Mol Genet Metab. 2005 Dec;86 Suppl 1:S54-60. doi: 10.1016/j.ymgme.2005.05.014. Epub 2005 Jul 22. PMID 16040265
- [Background] Kuvan® Package Insert. BioMarin. 2007
- [Background] Blau N. Defining tetrahydrobiopterin (BH4)-responsiveness in PKU. J Inherit Metab Dis. 2008 Feb;31(1):2-3. doi: 10.1007/s10545-007-9979-1. No abstract available. PMID 18327672
- [Background] Fiege B, Blau N. Assessment of tetrahydrobiopterin (BH4) responsiveness in phenylketonuria. J Pediatr. 2007 Jun;150(6):627-30. doi: 10.1016/j.jpeds.2007.02.017. PMID 17517248
- [Background] Levy H, Burton B, Cederbaum S, Scriver C. Recommendations for evaluation of responsiveness to tetrahydrobiopterin (BH(4)) in phenylketonuria and its use in treatment. Mol Genet Metab. 2007 Dec;92(4):287-91. doi: 10.1016/j.ymgme.2007.09.017. PMID 18036498
- [Background] Zurfluh MR, Zschocke J, Lindner M, Feillet F, Chery C, Burlina A, Stevens RC, Thony B, Blau N. Molecular genetics of tetrahydrobiopterin-responsive phenylalanine hydroxylase deficiency. Hum Mutat. 2008 Jan;29(1):167-75. doi: 10.1002/humu.20637. PMID 17935162
- [Background] Fernhoff P, Burton B, Nowacka M, Hennermann J, Kakkis E, Dorenbaum PKU-008: A Long-Term, Open-Label Study of Sapropterin Dihydrochloride (Kuvan®) in PKU Subjects. Poster at the 2009 American College of Medical Genetics Annual Clinical Genetics Meeting.
- [Background] Levy HL, Milanowski A, Chakrapani A, Cleary M, Lee P, Trefz FK, Whitley CB, Feillet F, Feigenbaum AS, Bebchuk JD, Christ-Schmidt H, Dorenbaum A; Sapropterin Research Group. Efficacy of sapropterin dihydrochloride (tetrahydrobiopterin, 6R-BH4) for reduction of phenylalanine concentration in patients with phenylketonuria: a phase III randomised placebo-controlled study. Lancet. 2007 Aug 11;370(9586):504-10. doi: 10.1016/S0140-6736(07)61234-3. PMID 17693179
- [Background] Trefz FK, Burton BK, Longo N, Casanova MM, Gruskin DJ, Dorenbaum A, Kakkis ED, Crombez EA, Grange DK, Harmatz P, Lipson MH, Milanowski A, Randolph LM, Vockley J, Whitley CB, Wolff JA, Bebchuk J, Christ-Schmidt H, Hennermann JB; Sapropterin Study Group. Efficacy of sapropterin dihydrochloride in increasing phenylalanine tolerance in children with phenylketonuria: a phase III, randomized, double-blind, placebo-controlled study. J Pediatr. 2009 May;154(5):700-7. doi: 10.1016/j.jpeds.2008.11.040. Epub 2009 Mar 4. PMID 19261295
- [Background] Luciana M, Sullivan J, Nelson CA. Associations between phenylalanine-to-tyrosine ratios and performance on tests of neuropsychological function in adolescents treated early and continuously for phenylketonuria. Child Dev. 2001 Nov-Dec;72(6):1637-52. doi: 10.1111/1467-8624.00370. PMID 11768137
- See also: Arnold GL. Phenylketonuria, Publication Link — http://emedicine.medscape.com/article/947781-overview

RESULTS

PARTICIPANT FLOW:
Groups:
- Kuvan®: Kuvan® (sapropterin dihydrochloride) oral solution 20 milligram per kilogram (mg/kg) once daily for 28 +/- 1 days.
Period: Overall Study
Arm/Group | Kuvan®
Started | 59
Completed | 58
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Kuvan®
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 30 Percent Reduction From Baseline in Blood Phenylalanine (Phe) Level
Description: Response to treatment was defined as 30 percent reduction from Baseline in blood phenylalanine (Phe) Level during the 28 +/- 1 days.
Time Frame: Baseline up to Day 28 +/- 1
Population: Full analysis set (FAS) population included all the participants with a valid Baseline blood Phe level measure and who received at least one dose of Kuvan®.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 59
Percentage of participants | 75 [62 to 85]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Treatment Emergent Adverse Events, Treatment Related Adverse Events and AEs Leading to Withdrawal
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Baseline up to Day 42 +/- 3
Population: Safety population included all the participants with a valid Baseline blood Phe level measure and who received at least one dose of Kuvan®.
Measure: Number; unit: Participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 59
Participants
  AEs | 58
  Treatment Emergent AEs | 57
  Treatment Related AEs | 36
  AEs leading to withdrawal | 1

3. Secondary Outcome: Percentage of Early-, Late-, Partial-Responders and Non-responders to Treatment With Kuvan®
Description: Early responders defined as percentage of participants with at least 30 percent reduction in Phe levels within the first seven days of treatment. Late responders defined as percentage of participants with less than 30 percent reduction in Phe levels within first seven days of treatment, but at least 30 percent reduction in Phe levels within 28 +/- 1 days of treatment. Partial responders defined as percentage of participants with Phe levels reduction between 10 and 30 percent at any blood measurement within the 28 +/- 1 days of treatment. Non-responders defined as percentage of participants with a Phe level reduction of less than 10 percent within 28 +/- 1 days.
Time Frame: Baseline up to Day 28 +/- 1
Population: FAS population included all the participants with a valid Baseline blood Phe level measure and who received at least one dose of Kuvan®.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 59
Percentage of participants
  Early Responders | 64.4 [50.9 to 76.4]
  Late Responders | 10.2 [3.8 to 20.8]
  Partial Responders | 25.4 [15.0 to 38.4]
  Non-responders | 0 [0 to 0]

4. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 30 Percent, 20 to 30 Percent, 10 to 20 Percent and Less Than (<) 10 Percent Reduction in Blood Phe Levels According to Phenylketonuria (PKU) Phenotypes
Description: The Phenylketonuria (PKU) is categorized as per phenotype into classical PKU: (blood Phe levels greater than [>] 1200 micromole per liter [mcmol/l]), mild PKU (blood Phe levels 600 to 1200 mcmol/l), mild Hyperphenylalaninaemia (HPA) (blood Phe levels 300 to 600 mcmol/l).
Time Frame: Baseline up to Day 28 +/- 1
Population: FAS population included all the participants with a valid Baseline blood Phe level measure and who received at least one dose of Kuvan®. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure. 'n' signifies number of participants who were evaluable for specified categories at different time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 55
Percentage of participants
  Mild HPA: >= 30 percent (n=7) | 57
  Mild HPA: 20 to 30 percent (n=7) | 29 (24.9)
  Mild HPA: 10 to 20 percent (n=7) | 0 (25.4)
  Mild HPA: < 10 percent (n=7) | 14 (33.4)
  Mild PKU: >= 30 percent (n=26) | 69 (96.2)
  Mild PKU: 20 to 30 percent (n=26) | 8 (64.9)
  Mild PKU: 10 to 20 percent (n=26) | 4 (60.8)
  Mild PKU: < 10 percent (n=26) | 19 (69.3)
  Classical PKU: >= 30 percent (n=22) | 45 (83.8)
  Classical PKU: 20 to 30 percent (n=22) | 0
  Classical PKU: 10 to 20 percent (n=22) | 23
  Classical PKU: < 10 percent (n=22) | 32

5. Secondary Outcome: Percentage of Early-, Late- and Partial-Responders According to Phenotype
Description: The PKU is categorized as per phenotype into classical PKU: (blood Phe levels > 1200 mcmol/l), mild PKU (blood Phe levels 600 to 1200 mcmol/l), mild HPA (blood Phe levels 300 to 600 mcmol/l). Early responders defined as percentage of participants with at least 30 percent reduction in Phe levels within the first seven days of treatment. Late responders defined as percentage of participants with less than 30 percent reduction in Phe levels within first seven days of treatment, but at least 30 percent reduction in Phe levels within 28 +/- 1 days of treatment. Partial responders defined as percentage of participants with Phe levels reduction between 10 and 30 percent at any blood measurement within the 28 +/- 1 days of treatment.
Time Frame: Baseline up to Day 28 +/- 1
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Kuvan®
Number analyzed (Participants) | 56
Percentage of participants
  Mild HPA: Early Responders (n=7) | 86
  Mild HPA: Late Responders (n=7) | 0
  Mild HPA: Partial Responders (n=7) | 14
  Mild PKU: Early Responders (n=26) | 85
  Mild PKU: Late Responders (n=26) | 4
  Mild PKU: Partial Responders (n=26) | 12
  Classical PKU: Early Responders (n=23) | 39
  Classical PKU: Late Responders (n=23) | 17
  Classical PKU: Partial Responders (n=23) | 43

6. Secondary Outcome: Mean Change From Baseline in Blood Phenylalanine-to-tyrosine Ratio
Description: Phenylalanine-to-tyrosine ratio is the best indicator of dopamine availability in PKU. The change in blood phenylalanine-to-tyrosine ratio at Day 28 was calculated as blood phenylalanine-to-tyrosine ratio at Day 28 minus blood phenylalanine-to-tyrosine ratio at Baseline.
Time Frame: Baseline, Day 28
Population: FAS population included all the participants with a valid Baseline blood Phe level measure and who received at least one dose of Kuvan®. 'n' signifies number of participants who were evaluable for specified categories at different time points.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Kuvan®
Number analyzed (Participants) | 59
Ratio
  Baseline (n=59) | 10.978 (5.978)
  Change at Day 28 (n=58) | -2.136 (3.948)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 42 +/- 3
Description: An adverse event is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Kuvan®
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 58/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan® (N=59)
Dizziness (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 2
Eye pruritus (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 6
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastroenteritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival pruritus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Oropharyngeal pain (Gastrointestinal disorders) | 2
Tongue blistering (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Discomfort (General disorders) | 1
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 3
Listless (General disorders) | 1
Malaise (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 5
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Injury (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Amino acid level decreased (Investigations) | 21
Decreased appetite (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint lock (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 25
Migraine (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Irritability (Psychiatric disorders) | 1
Somatoform disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 4
Acute tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Migraine (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other